CLINICAL TRIAL: NCT00579618
Title: Ascertainment of Saliva or Blood Samples For Genetic Epidemiology Studies of Cancer and Aging
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Beth Abraham (Unknown); Gurwin Jewish Nursing & Rehabilitation Center (Other); Hebrew Home at Riverdale (Other); Jewish Home & Hospital Lifecare System (Other); Margaret Tietz Nursing and Rehabilitation Center (Other); Metropolitan Jewish Health System (Other); Northern Services Group (Unknown); Parker Jewish Institute (Unknown); Lenox Hill Neighborhood House (Other); JASA at Temple Emanuel of Parkchester Senior Center (Unknown); Van Cortlandt Village Senior Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-102
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Non-cancer Affected Volunteers
Keywords: non-cancer affected volunteers; aged 60 years or older
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva or blood samples

INTERVENTIONS:
Other: Saliva or Blood samples — Extracting sample of saliva or blood only once.

SUMMARY:
The purpose of this study is to help us learn more about the roles of genes in cancers. Genes are short pieces of DNA which determine the inherited characteristics that distinguish one individual from another. This study will look at how some genes might raise or lower the chance some people may develop cancer. The sample collection will help generate the materials needed for this study.

DETAILED DESCRIPTION:
This is a protocol to obtain saliva or blood samples from non-cancer affected volunteers aged 60 years or older, without a history of cancer other than non-melanoma skin cancer. These samples will be used in a genomic approach to elucidate novel pathways of cancer predisposition.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must be non-cancer affected volunteers of either gender who are 60 years of age or older at the time of saliva/blood donation.
* Subjects will self-identify religion and country of origin of grandparents.
* Volunteers will have (by self report) no history of cancer other than nonmelanoma skin cancer. It is recognized that there may be some errors in self report, however, the literature reports a very low error rate for self reported disease reporting for cancer as assessed by interview.

Exclusion Criteria:

* Subjects with mental impairment will be excluded from this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing homes, senior centers, health fairs or other community organizations.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
obtain saliva or blood from non-cancer volunteers, 60 years or older to carry out anonymous genetic epidemiology studies related to resistance to cancer in elderly. | conclusion of the study

SECONDARY OUTCOMES:
samples perform high density genomic scans & candid gene studies carriers specif BRCA found mutat who haven't been affect by breast cancer & old than 60 find genetic cofactor may modify a predispo breast ca confer by germline mutation in BRCA1 & BRCA2. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Web Site — http://www.mskcc.org